CLINICAL TRIAL: NCT01480713
Title: Impact of Raltegravir Intensification on HIV-1-infected Subjects With Complete Viral Suppression Under Monotherapy With Protease Inhibitors. A 24-week Open-label, Proof-of-concept Pilot Clinical Trial.
Brief Title: Impact of Raltegravir Intensification on HIV-1-infected Subjects With Complete Viral Suppression Under Monotherapy With Protease Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IrsiCaixa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIPIM; 2011-004464-30
Record Dates: First submitted 2011-11-21; First posted 2011-11-29 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: HIV-1 Infection
Keywords: HIV-1; protease inhibitors; integrase inhibitors; raltegravir; viral replication; treatment intensification; viral pathogenesis; immune activation
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monotherapy with IPs+ Raltegravir 400 mg (Experimental): Lopinavir/r 400/100 mg every 12 hours + Raltegravir 400 mg every 12 hours or Darunavir/rit 800/100 mg every 24 hours + Raltegravir 400 mg every 12 hours
  Interventions: Drug: Isentress® (Raltegravir, 400 mg every 12 hours); Drug: Isentress® (Raltegravir, 400 every 12 hours)

INTERVENTIONS:
Drug: Isentress® (Raltegravir, 400 mg every 12 hours) — Lopinavir/r 200/50 mg every 12 hours + Raltegravir 400 mg every 12 hours
  Other Names: N/H
Drug: Isentress® (Raltegravir, 400 every 12 hours) — Darunavir/rit 800/100 mg every 24 hours + Raltegravir 400 mg every 12 hours
  Other Names: N/H

SUMMARY:
This is a pilot, proof of concept, open-label clinical trial, to assess the extend of persistent viral reservoir and the level of immune activation in patients receiving suppressive treatment with protease inhibitors.

40 Chronically HIV-1 infected subjects, receiving monotherapy with ritonavir-boosted lopinavir or darunavir for at least 12 months with plasma viremia below 50 copies HIV RNA per ml, and CD4 T-cell counts greater than 500 cells/mm3 will be included.

The total duration of the study will be 48 weeks: 12 weeks for patients' inclusion, 24 weeks of follow-up once the last patient is included, and 12 weeks for data analysis.

DETAILED DESCRIPTION:
AIDS continues to be a major global health priority. Although important progress has been achieved in preventing new HIV infections and in lowering the annual number of AIDS-related deaths, the number of people living with HIV worldwide continued to grow in 2008, reaching an estimated 33.4 million. AIDS-related illnesses remain one of the leading causes of death globally and are projected to continue as a significant global cause of premature mortality in the coming decades: an estimated 3 million new HIV infections and 2 million deaths due to AIDS-related illnesses occurred worldwide in 2008 (UNAIDS, report 2009).

In contrast to the failed attempts at developing a vaccine against HIV, efforts to provide drug therapies stand as a great success. More than 25 agents have been approved thus far, and the right combinations can suppress replication of the virus, often keeping blood levels so low as to be undetectable by standard tests. These powerful drug combinations, collectively termed highly active antiretroviral therapy, HAART, have prolonged life and health in countless infected individuals.

Although life expectancy of HAART-treated people in developed countries has significantly improved, treatment has to be carefully observed to avoid virus rebound, what will happen in only in a few days after treatment withdrawal (13). Moreover, long-term treatment is not exempt from complications, including the continuous likelihood of developing drug resistance and the induction of significant metabolic disturbances as a consequence of drug toxicities, which will clinically impact on the future health of the HIV-infected patient, including hyperlipidaemia, lipodystrophy, metabolic syndrome, cardiovascular disease and type 2 diabetes. Finally, the cost of full HIV-1 treatment implementation should not be disregarded. Only in Catalunya, the annual cost in antiretroviral approaches the 300 million Euros.

Guidelines for the use of antiretrovirals for HIV-1 infection recommend combining at least three agents. However, toxicities, cost, and the complexity of such regimens warrant the search for other options. Boosted protease inhibitor monotherapy is one of the appealing options being investigated.

Different clinical trials have evaluated the efficacy of boosted protease inhibitor monotherapy in several clinical settings: maintenance therapy of HAART-suppressed subjects (1-3, 12), salvage regimens (10) and first-line treatment (4, 7-9). Monotherapies with boosted lopinavir or darunavir have been largely investigated in maintenance and induction-maintenance strategies, showing that they are able to maintain viral suppression in a high proportion of patients. Thus, both Darunavir/ritonavir DRV/r and Lopinavir/ritonavir LPV/r are accepted options for monotherapy regimens when triple therapy is not possible.

To determine the role for low-level replication in maintaining HIV infection, our group has recently exploited the unique effect of Raltegravir on viral replication (6). This integrase inhibitor blocks integration of viral linear cDNA into genomic host cell DNA. Under normal conditions, in the absence of raltegravir, a small proportion of the linear cDNA is circularized by host DNA repair enzymes to form episomes with one or two copies of the viral long terminal repeat(LTR)(1-LTR or 2-LTR circles). We reasoned that if there was persistent, ongoing low-level viral replication in patients on antiretroviral therapy, raltegravir administration should result in a measurable increase in 2-LTR circles in their blood, as happened. Furthermore, the 2-LTR-positive subjects receiving raltegravir showed marked decreases in CD8+ T-cell activation markers, providing what may be the first in vivo demonstration that ongoing immune activation is attributable, in part, to ongoing, albeit low-level, viral replication.

It seems likely that the contribution of each mechanism to maintaining HIV infection varies from person to person and is dependent on multiple variables, including genetics, development of resistance, concurrent infections, viral strain, stage of disease and antiretroviral regimen. In fact, among patients receiving raltegravir in the study, the main difference between the 2-LTR-positive and 2-LTR-negative groups was the antiretroviral regimen used: a total of 61% of patients in the 2-LTR-positive group was on a protease inhibitor-containing regimen at the time raltegravir was added, compared to 19% of the 2-LTR-negative group (P = 0.011). It is possible that the presence of three reverse transcriptase inhibitors in protease inhibitor-sparing regimens reduces the probability of formation of the linear cDNA precursor to episomal cDNA. It is also possible that active replication occurs in anatomic compartments that are less accessible to protease inhibitors or that pharmacodynamic variability of protease inhibitors contributes to this observation.

To further explore the previous observations, we have designed a pilot trial in which patients that have been on boosted protease inhibitor single-agent strategy with suppressive plasma viremia by standard assays would have their treatment temporary intensified with raltegravir. This should provide further insights in the level of residual viral replication and immune-affectation of patients on boosted protease inhibitor monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults (≥18 years old).
2. Absence of prior virological failure with protease inhibitors (PIs).
3. No mono or dual protease inhibitor therapy previous to HAART initiation.
4. Patients had to be on monotherapy with ritonavir-boosted lopinavir (LPV/r 400/100 mg every 12 hours) or darunavir (DRV/r 800/100 mg every 24 hours) for ≥ 12 months. Switching from standard HAART to protease inhibitor monotherapy had to happen with undetectable plasma viremia.
5. Complete virological suppression (<50 copies/mL) for ≥12 months, including at least 2 times during the last year.
6. CD4 cell count ≥500 cells/µL.
7. Availability (if possible, not mandatory) of a genotype prior to the start of HAART, with absence of any major drug-related mutations.
8. Voluntary written informed consent.

Exclusion Criteria:

1. Lactating, pregnancy, or fertile women willing to be pregnant.
2. Active substance abuse or major psychiatric disease.
3. Presence of any polymorphism or mutation associated to raltegravir resistance at baseline (prior to first HAART).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from week -8 in Integrated viral HIV-1 DNA in A peripheral blood mononuclear cells (PBMCs) at 8 months. | week -8, -4, Baseline, week 4, 12 and 24
Change from week -8 in Unintegrated viral HIV-1 DNA in PBMCs at 8 months. | week -8, -4, Baseline, week 1, 2, 4, 8, 12 and 24
Change from week -8 in lymphocyte activation markers in PBMCs at 8 months. | week -8, -4, Baseline, week 4, 8, 12 and 24

SECONDARY OUTCOMES:
ultrasensitive HIV-1 viral load | week -8, -4, Baseline, week 1, 2, 4, 8, 12 and 24
viral load >50 copies/mL | week -8, -4, Baseline, week 1, 2, 4, 8, 12 and 24
HIV-1 RNA below 50 copies/mL. | week 24 and 48
Change in the lymphocyte activation markers | week -8, -4, Baseline, week 1, 2, 4, 8, 12, and 24 and 48.
Change in the inflammation markers (soluble CD14, IL-6, D-Dimer, vCam, C Reactive Protein) | week -8, -4, Baseline, week 4, 8, 12, and 24 and 48

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Puertas MC, Gomez-Mora E, Santos JR, Molto J, Urrea V, Moron-Lopez S, Hernandez-Rodriguez A, Marfil S, Martinez-Bonet M, Matas L, Munoz-Fernandez MA, Clotet B, Blanco J, Martinez-Picado J. Impact of intensification with raltegravir on HIV-1-infected individuals receiving monotherapy with boosted PIs. J Antimicrob Chemother. 2018 Jul 1;73(7):1940-1948. doi: 10.1093/jac/dky106. PMID 29635527